CLINICAL TRIAL: NCT04340531
Title: Break Free: Effectiveness of a Multi-Level Smoking Cessation Program Adapted for High-Risk Women in Rural Communities
Brief Title: Effectiveness of a Multi-Level Smoking Cessation Program for High-Risk Women in Rural Communities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Amy Ferketich, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-20056; NCI-2020-01403 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA229143 (NIH)
Record Dates: First submitted 2020-03-24; First posted 2020-04-09 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-04

CONDITIONS: Tobacco-Related Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (early arm) (Experimental): Providers undergo training over 60 minutes to explain the Break Free program and basics of quitting smoking during months 13-24. Female smokers interested in quitting in the next 6 months will be referred to an in-person counseling session at the clinic. Participants then receive 4 phone counseling over 15-20 minutes with a trained tobacco treatment specialist.
  Interventions: Other: Survey Administration; Other: Tobacco Cessation Counseling; Other: Training
- Arm II (delayed arm) (Active Comparator): Female smokers receive usual care during months 13-24. Providers undergo training over 60 minutes to explain the Break Free program and basics of quitting smoking during months 25-36. Female smokers interested in quitting in the next 6 months will be referred to an in-person counseling session at the clinic. Participants then receive 4 phone counseling over 15-20 minutes with a trained tobacco treatment specialist.
  Interventions: Other: Best Practice; Other: Survey Administration; Other: Tobacco Cessation Counseling; Other: Training

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (delayed arm)
Other: Survey Administration — Ancillary studies
Other: Tobacco Cessation Counseling — Receive referred to counseling session
Other: Tobacco Cessation Counseling — Receive phone counseling
Other: Training — Undergo training
  Other Names: Training Programs

SUMMARY:
This phase IV trial examines the effectiveness of a multi-level smoking cessation program for high-risk women in rural communities. Cigarette smoking is a major risk factor for cervical cancer in women. Rural primary care practices and providers often lack the electronic health record support to pre-identify smokers for services, as well as lack the necessary counseling training and access to comprehensive cessation programs. Implementing evidence-based smoking cessation programs in rural Appalachia may decrease the rates of cigarette smoking and as a result decrease the rates of cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effectiveness of a core component of an integrated cervical cancer prevention program designed to help female smokers quit by standardizing clinical practice supports and protocols. (Service outcomes) II. Determine satisfaction with the multilevel intervention. (Client outcomes) III. Test the sustainability of the multilevel intervention via training of providers and staff on counseling and billing for evidence-based smoking cessation services. (Implementation outcomes)

OUTLINE:

IMPLEMENTATION OF TOBACCO-USER IDENTIFICATION SYSTEM: Clinics and systems develop and implement minimally required electronic tracking and reporting systems for identification of smokers during months 1-12.

GROUP RANDOMIZED TRIAL: Providers and participants are randomized to 1 of 2 arms.

ARM I (EARLY ARM): Providers undergo training over 60 minutes to explain the Break Free program and basics of quitting smoking during months 13-24. Female smokers interested in quitting in the next 6 months will be referred to an in-person counseling session at the clinic. Participants then receive 4 phone counseling over 15-20 minutes with a trained tobacco treatment specialist.

ARM II (DELAYED ARM): Female smokers receive usual care during months 13-24. Providers undergo training over 60 minutes to explain the Break Free program and basics of quitting smoking during months 25-36. Female smokers interested in quitting in the next 6 months will be referred to an in-person counseling session at the clinic. Participants then receive 4 phone counseling over 15-20 minutes with a trained tobacco treatment specialist.

ELIGIBILITY:
Inclusion Criteria:

* HEALTH SYSTEM/CLINIC
* Based in one of the Appalachian regions included in this program project
* Provides care to female smokers
* PROVIDER
* Practicing in one of the participating health systems
* Involved in patient care
* PATIENT
* Females
* Age 18 to 64
* Smokers who consume at least 5 cigarettes per day (less than the minimum in most cessation studies, yet still enough to show signs of nicotine dependence)
* Ready to quit smoking in the next 6 months
* English-speaking
* Able to participate in counseling
* Willing to try smoking cessation pharmacotherapy
* Not pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 810 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of intervention - delivery of AAC | Up to 6 months
  This provider-level outcome includes self-reported changes in the delivery of the Ask, Advise, and Connect (AAC).
Acceptability of intervention - referral rate | Up to 6 months
  This provider-level outcome includes the rate of referrals to the in-clinic smoking cessation counselor.
Fidelity to the intervention: counseling calls | Day after phone counseling during the span of the intervention (one year)
  Measured by asking 10% of randomly selected women questions about content of the phone counseling.
Fidelity to the intervention: provider visits | At time of in person visit for a one week span, every other month during the span of the intervention (one year)
  Measured by self-administered, anonymous, post-provider visit surveys every other month by patients who were in the clinic for a visit during a one-week period. Patients will be asking whether the provider asked about tobacco use, if a smoker, advised the patient to quit, discussed cessation, and connected the smoker to counseling.
Sustainability of the intervention: clinic continuation of Break Free | During the span of the final phase of study (2 years)
  Measured by self-reported continuation of cessation counseling by clinic staff
Sustainability of the intervention: counseling sessions | During the span of the final phase of study (2 years)
  Measured by the number of counseling sessions billed for overall
Sustainability of the intervention: counseling sessions per smoker | During the span of the final phase of study (2 years)
  Measured by the number of counseling sessions billed for each individual smoker who has at least one session
Sustainability of the intervention: EHR documentation | During the span of the final phase of study (2 years)
  Measured by electronic health record documentation of tobacco use
Cost-effectiveness of intervention | Up to 6 months
  Will be assessed using standard costs by considering costs of each component including pharmacotherapy, clinic counselor time and training, smoking cessation counselor time and training, telephone and material costs, and other administrative costs.
Effectiveness of intervention at increasing brief cessation counseling: Change over time | 3 months, 6 months, 12 months
  Will be assessed using patient post-visit surveys and see if they increase over time.
Point prevalence | Up to 7 days
  Measured using self-report of any tobacco use. Abstainers will be classified as those participants who self-report no use of tobacco during the past week.
Floating abstinence | Up to 7 days
  Defined as not smoking during any consecutive 7-day period since the last assessment. Self-reported by patients.
Prolonged abstinence | At each follow-up visit over the span of the intervention (1 year)
  Defined as no smoking after a two-week grace period from the quit date. Self-reported by patients.
Provider satisfaction | Mid-points of each provider arm during the intervention year (1 year)
  Measured via provider surveys
Staff satisfaction | Mid-points of each provider arm during the intervention year (1 year)
  Measured via staff surveys
Smoker satisfaction with Break Free counseling | At the end of each Break Free counseling sessions during the intervention year (year 1)
  Measured via patient surveys
Smoker satisfaction during Break Free counseling | At the end of each Break Free counseling sessions during the intervention year (year 1)
  Measured via patient surveys
Smoker satisfaction after Break Free program | At 6 months after completion of Break Free counseling
  Measured via patient surveys
Change in provider knowledge | Baseline, post-training (same day), 1 year
  Using the Theory of Planned Behavior (TPB) model, effectiveness of intervention on improved provider knowledge will be assessed.
Change in provider attitudes | Baseline, post-training (1 day), 1 year
  Using the Theory of Planned Behavior (TPB) model, effectiveness of intervention on improved provider attitudes will be assessed.
Change in provider's normative beliefs | Baseline, post-training (1 day), 1 year
  Using the Theory of Planned Behavior (TPB) model, effectiveness of intervention on provider's normative beliefs will be assessed.
Change in provider's perceived behavioral control | Baseline, post-training (1 day), 1 year
  Using the Theory of Planned Behavior (TPB) model, effectiveness of intervention on provider's perceived behavioral control will be assessed.
Effectiveness of intervention of Improved provider knowledge and attitude | Baseline, post-training (1 day), 1 year
  Using the Theory of Planned Behavior (TPB) model, attitudes, normative beliefs, and perceived behavioral control will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Ferketich, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (4):
- United States (4):
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patterson JG, Borger TN, Burris JL, Conaway M, Klesges R, Ashcraft A, Hauser L, Clark C, Wright L, Cooper S, Smith MC, Dignan M, Kennedy-Rea S, Paskett ED, Anderson R, Ferketich AK. A cluster randomized controlled trial for a multi-level, clinic-based smoking cessation program with women in Appalachian communities: study protocol for the "Break Free" program. Addict Sci Clin Pract. 2022 Feb 14;17(1):11. doi: 10.1186/s13722-022-00295-5. PMID 35164857
- See also: The Jamesline — http://cancer.osu.edu